CLINICAL TRIAL: NCT06157372
Title: Detection of Pathogen and Antibiotic Resistance Genes by Targeted Next-Generation Sequencing Compared With Metagenomic Next-Generation Sequencing in ICU Patients.
Brief Title: Detection of Pathogen and Antibiotic Resistance Genes by Targeted Next-Generation Sequencing in ICU Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-667-03
Record Dates: First submitted 2023-10-19; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Infections; Critical Illness; Diagnosis
Keywords: Targeted Next-generation sequencing; ICU; infections; Next-generation sequencing
MeSH Terms: conditions — Infections; Critical Illness; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and qualified lower respiratory tract specimens (LRS), including bronchoalveolar lavage fluid (BALF), pleural/peritoneal effusion, lymph node tissue and other suspected infected tissues are obtained from patients after including and preferred to be collected before the antimicrobial therapy began.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Infection group: Participants received traditional etiological culture of suspected site of infection.
  Interventions: Diagnostic Test: targeted next-generation sequencing (tNGS)
- Infection group: Participants received traditional etiological culture, metagenomic next-generation sequencing of infectious sites.
  Interventions: Diagnostic Test: targeted next-generation sequencing (tNGS)

INTERVENTIONS:
Diagnostic Test: targeted next-generation sequencing (tNGS) — To provide rapid etiological diagnosis of patients by means of targeted next-generation sequencing.

SUMMARY:
It is difficult to determine the pathogens in the early stage of infection in critically ill patients, and empirical use of broad-spectrum antibiotics for a long time is often necessary, leading to antibiotics drug resistance. Targeted next generation sequencing (tNGS) can provide faster results for pathogen and related antibiotic resistant diagnosis. But it lacks sufficient clinical evidence. Evidence regarding the clinical diagnostic accuracy and drug resistance is needed to comprehensively evaluate targeted next generation sequencing (tNGS) for diagnosis of patients in ICU who and will be critical to inform national policy.

DETAILED DESCRIPTION:
Infectious diseases are one of the highest mortality and morbidity diseases in humans. Due to the difficulty in identifying the pathogen in the early stage of infection, patients with severe infections often need to empirically use broad-spectrum antimicrobials for a long time. The traditional gold standard of etiological detection - etiological culture, even in sepsis patients, only about 60% of the results are positive. Therefore, the accurate identification and rapid classification of pathogenic microorganisms is very important for the patient's precise diagnosis and timely treatment.

Metagenomic next generation sequencing (mNGS), which has emerged in recent years, have been shown to provide early diagnosis and targeted medication guidance for bloodstream infections and respiratory infections, but it is expensive and not able to provide related drug resistant genes. Therefore, targeted next generation sequencing (tNGS) has been derived, which is characterized by rapid sequencing and genetic testing for drug resistance.

The purpose of this study is to evaluate the efficacy of etiological diagnosis and provide patients with more accurate treatment.

ELIGIBILITY:
Inclusion Criteria:

* The presence of an infection or clearly excluded the presence of infection.
* Etiological culture and/or metagenomic next-generation sequencing detection of specimens sent for testing.

Exclusion Criteria:

* Suspected infection.
* Participation in other clinical trials in the past 2 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in ICU truly have infected disease and non-infected disease diagnosed by two ICU physicians determining whether the patient have an infectious etiology and identifying the pathogen through existing clinical guidelines, clinical features, laboratory tests, microbiological tests, chest imaging, and treatment response.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 year
  The probability of being positive in clinical composite diagnosis, the probability that etiological culture, mNGS, and tNGS tests are also positive, which is also known as the true positive rate.
Specificity | 1 year
  It refers to the probability that cultures, mNGS, and tNGS tests are also negative in the presence of non-infection confirmed by the gold standard.

SECONDARY OUTCOMES:
False-positive rate | 1 year
  It refers to the probability that the gold-standard confirmed absence of infection is also positive for etiological culture, mNGS, and tNGS tests.
False-negative rate | 1 year
  It refers to the probability of being positive in the clinical composite diagnosis, and the probability that etiological cultures, mNGS, and tNGS tests will also be negative.
Positive predictive value | 1 year
  Positive predictive value is the probability that subjects with a positive test truly have the disease.
Negative predictive value | 1 year
  Negative predictive value is the probability that subjects with a negative screening test truly don't have the disease.
Kappa values | 1 year
  Kappa values are used to measure the agreement between two raters. The range of possible values of kappa is from -1 to 1, though it usually falls between 0 and 1. Unity represents perfect agreement, indicating that the raters agree in their classification of every case. Kappa values of 0.41~0.60 are moderately consistent, 0.61~0.80 are basically consistent, and 0.81~1.00 is almost identical.
Drug resistant gene by targeted next-generation sequencing | 1 year
  It refers to the distribution of drug resistance by targeted next-generation sequencing using the Comprehensive Antibiotic Resistance Database.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijie He, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu CY, Miller SA. Clinical metagenomics. Nat Rev Genet. 2019 Jun;20(6):341-355. doi: 10.1038/s41576-019-0113-7. PMID 30918369
- [Background] Diao Z, Han D, Zhang R, Li J. Metagenomics next-generation sequencing tests take the stage in the diagnosis of lower respiratory tract infections. J Adv Res. 2021 Sep 29;38:201-212. doi: 10.1016/j.jare.2021.09.012. eCollection 2022 May. PMID 35572406
- [Background] Miao Q, Ma Y, Wang Q, Pan J, Zhang Y, Jin W, Yao Y, Su Y, Huang Y, Wang M, Li B, Li H, Zhou C, Li C, Ye M, Xu X, Li Y, Hu B. Microbiological Diagnostic Performance of Metagenomic Next-generation Sequencing When Applied to Clinical Practice. Clin Infect Dis. 2018 Nov 13;67(suppl_2):S231-S240. doi: 10.1093/cid/ciy693. PMID 30423048
- [Background] Pei XM, Yeung MHY, Wong ANN, Tsang HF, Yu ACS, Yim AKY, Wong SCC. Targeted Sequencing Approach and Its Clinical Applications for the Molecular Diagnosis of Human Diseases. Cells. 2023 Feb 2;12(3):493. doi: 10.3390/cells12030493. PMID 36766834
- [Background] Li S, Tong J, Liu Y, Shen W, Hu P. Targeted next generation sequencing is comparable with metagenomic next generation sequencing in adults with pneumonia for pathogenic microorganism detection. J Infect. 2022 Nov;85(5):e127-e129. doi: 10.1016/j.jinf.2022.08.022. Epub 2022 Aug 26. No abstract available. PMID 36031154
- [Background] Gaston DC, Miller HB, Fissel JA, Jacobs E, Gough E, Wu J, Klein EY, Carroll KC, Simner PJ. Evaluation of Metagenomic and Targeted Next-Generation Sequencing Workflows for Detection of Respiratory Pathogens from Bronchoalveolar Lavage Fluid Specimens. J Clin Microbiol. 2022 Jul 20;60(7):e0052622. doi: 10.1128/jcm.00526-22. Epub 2022 Jun 13. PMID 35695488